CLINICAL TRIAL: NCT06073405
Title: MEasuring the Accuracy of an Artificial Intelligence Tool That Establishes Polyp Size in Real-time
Brief Title: Colonic Polyp Size Measurement With Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giulio Antonelli, Principal Investigator, University of Roma La Sapienza
Other Study IDs: METER
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Colon Polyp; Artificial Intelligence
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Colonic Polyp Measurement Assessment Via Artificial Intelligence — In this study, we collect colonoscopy video clips of polyps and, among the related clinical information, their estimated size using the gold standard technique, and we use them offline to evaluate the measurement performances of the novel virtual polyp sizing tool

SUMMARY:
Primary objective of the study is to evaluate if the novel virtual polyp sizing tool accuracy in determining the size class of polyps among diminutive (0-5 mm), small (6-9 mm) and large (10 mm and above).

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 years or older undergoing colonoscopy
* Ability to provide written, informed consent (approved by EC) and understand the responsibilities of trial participation.

Exclusion criteria:

* Patients with known contra-indications to colonoscopy
* Patients who perform an emergency colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy for categorical distribution of polyp size | at study completion (this outcome is not an outcome measured from Time A to Time B but an outcome measured in one time point for all the colonoscopies performed in the study.
  1. Accuracy of the novel virtual polyp sizing tool in the determination of polyp size class among diminutive (0-5 mm), small (6-9 mm) and large (10 mm and above) as compared to the size estimated in-vivo by performing endoscopists with the help of a side-by-side forceps of known size

SECONDARY OUTCOMES:
Accuracy for continous determination of polyp size | at study completion (this outcome is not an outcome measured from Time A to Time B but an outcome measured in one time point for all the colonoscopies performed in the study.
  1. Polyp size in mm as determined by the novel virtual polyp sizing tool as compared to the size estimated in-vivo by performing endoscopists with the help of a side-by-side forceps of known size

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale dei Castelli, Ariccia, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes